CLINICAL TRIAL: NCT05687630
Title: Effect of Technology-assisted Physical Therapy for Patient With High Risk of Sarcopenia
Acronym: HRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202207113RINB
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-08

CONDITIONS: Sarcopenia
Keywords: sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-assisted group (Experimental)
  Interventions: Other: elastic band resisted exercise
- Traditional group (Active Comparator)
  Interventions: Other: elastic band resisted exercise

INTERVENTIONS:
Other: elastic band resisted exercise — muscle strengthening exercise, 10-15 times of each set, for 3 sets
  Other Names: resisted exercise

SUMMARY:
This research aims to identify whether the effects of video-assisted physical therapy, including home resistance training, is superior to traditional physical therapy, education leaflet for example.

This is an interventional research, single-blind, randomized control trail. We recruit high risk of sarcopenia people (low muscle strength and low physical performance) Two groups of participants are divided into traditional group and video-assisted group, both group are taught the same resisted exercise by physical therapist.

DETAILED DESCRIPTION:
Both group will record his/her baseline activity level with a given pedometer. After one week recording, we started initial evaluation (history taking, physical examination) and intervention.

Participants are taught thera-band resisted exercise, including large musculature of upper and lower extremities, each exercise are conducted 10-15 times for 3 sets.

Traditional group will receive an education leaflet and a notebook to record his/ her daily activity and frequency of exercise to record the compliance.

Video-assisted group will receive a QR code, which contain a website of exercise video on the cloud.

After 3 months intervention, participant will come back to our center for final examination.

ELIGIBILITY:
Inclusion Criteria:

* Age above 65 years old
* MMSE > 24 points
* walking more than 6 meters independently

Exclusion Criteria:

* people who cannot participate for 3 -day exercise for each week

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Grip strength | three months after initial evaluation
  use hand dynamometer to test maximal strength
walking speed | three months after initial evaluation
  walk for 4 meters to test the time that participant used
Timed up-and-go test | three months after initial evaluation

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | three months after initial evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu Kuo, Bachelor, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No